CLINICAL TRIAL: NCT00000843
Title: A Phase IA Single Dose Pharmacokinetics and Safety Study of the Oral Antiviral Compound, 9-[2-(Bispivaloyloxymethyl)Phosphonylmethoxyethyl]Adenine (Bis-POM PMEA) (Adefovir Dipivoxil) in Children With HIV-1 Infection
Brief Title: The Safety and Effectiveness of Adefovir Dipivoxil in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 310
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-04

CONDITIONS: HIV Infections
Keywords: Antiviral Agents; Adenine
MeSH Terms: conditions — HIV Infections | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
To evaluate the single-dose pharmacokinetic profile and acute toxicity of bis-POM PMEA ( adefovir dipivoxil ) in HIV-1 infected children, and to determine whether age-related differences exist. To ascertain dosages that may be suitable for a multiple-dose evaluation in this patient population.

Although the oral bioavailability of PMEA ( adefovir ) is low, the prodrug bis-POM PMEA has resulted in increased bioavailability in adult patients in clinical trials. However, the safety and pharmacokinetic patterns of drugs in infants often differ from those of adults and the direction of the variation is not predictable. This study will assess these parameters of bis-POM PMEA in children.

DETAILED DESCRIPTION:
Although the oral bioavailability of PMEA ( adefovir ) is low, the prodrug bis-POM PMEA has resulted in increased bioavailability in adult patients in clinical trials. However, the safety and pharmacokinetic patterns of drugs in infants often differ from those of adults and the direction of the variation is not predictable. This study will assess these parameters of bis-POM PMEA in children.

Patients are stratified by age, and separate cohorts from each age group receive 1 of 2 single doses of bis-POM PMEA. The lower dose is given to patients ages 3 months through 17 years; if toxicity is acceptable, the other cohort in this age range receives the higher dose. At this point, accrual of infants < 3 months old may begin at the lower dose, followed by accrual of this age group at the higher dose if toxicity is acceptable. Serum drug concentrations are monitored up to 8 hours post dose.

AS PER AMENDMENT 5/2/97: Based on data from both the low- and high-dose cohorts of the older age group (>= 3 months to < 18 years), the younger age group (<3 months) will be started at the high-dose.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Asymptomatic or mildly symptomatic HIV infection, with no worse than grade 1 toxicity for any symptoms.
* Consent of parent or guardian.

Prior Medication:

Allowed:

* IV gammaglobulin and aerosolized pentamidine for PCP prophylaxis.
* Antiretrovirals if discontinued by 72 hr prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Acute or chronic infections that require treatment during study.

Concurrent Medication:

Excluded:

* Antiretrovirals other than study drug.
* Other investigational agents.
* Immunomodulators.
* HIV-1 vaccines.
* Glucocorticoids.
* Drugs with potential for adverse interaction with study drug or that would interfere with quantitation of study drug in serum or plasma.
* TMP / SMX and dapsone.

PER AMENDMENT 8/23/96:

* Drugs which may affect renal excretion:
* Probenecid, Acyclovir, Ganciclovir, Foscarnet, Amphotericin B and Pentamidine.

Prior Medication:

Excluded within 72 hr prior to study entry:

* Antiretrovirals other than study drug.
* Other investigational agents.
* Immunomodulators.
* HIV-1 vaccines.
* Glucocorticoids.
* Drugs with potential for adverse interaction with study drug or that would interfere with quantitation of study drug in serum or plasma.
* TMP / SMX and dapsone.

PER AMENDMENT 8/23/96:

* Drugs which may affect renal excretion:
* Probenecid, Acyclovir, Ganciclovir, Foscarnet, Amphotericin B and Pentamidine.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: Hughes W, Study Chair; Shenep J, Study Chair
Locations (10):
- United States (9):
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173